CLINICAL TRIAL: NCT06833359
Title: Adaptation, Translation, and Cross-cultural Validation of the Cervical Disability Index (NDI) for Use in the Albanian-speaking Population
Brief Title: Validity, Reliability of Neck Disability Index in Albanian
Acronym: NDI
Status: Completed | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Jasemin Todri, Professor, Universidad Católica San Antonio de Murcia
Other Study IDs: 208/9
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Myofascial Pain Dysfunction Syndrome; Trigger Point Pain, Myofascial
Keywords: Validity; cross-cultural adaptation; Albanian Neck Disability index; Translation
MeSH Terms: conditions — Fibromyalgia; Myofascial Pain Syndromes | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — The Cervical Disability Index will be taught individually online through the Google questionnaire.

SUMMARY:
To translate and validate the Cervical Disability Index (NDI) into Albanian for use in the Albanian-speaking population

DETAILED DESCRIPTION:
The cross-cultural adaptation will be carried out according to the internationally recommended methodology, following the guidelines: translation, back-translation; dissemination of questionnaires and data collection and analysis.

Psychometric properties will be assessed by administering the questionnaire to approximately 400 participants. Reliability will be estimated by assessing stability and homogeneity.

ELIGIBILITY:
Inclusion Criteria:

* Myofascial syndrome
* Headache
* muscular pain
* articular pain
* arthirtis

Exclusion Criteria:

* contraindications to manual therapy
* severe trauma
* tumor
* metabolic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults with cervical pain
Sampling Method: Probability Sample
Enrollment: 582 (Actual)
Dates: Start 2025-02-16 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Albanian Neck Disability Index | 7 days
  An online questionnaire used to assess the impact of neck pain on patients' activities of daily living and quality of life which consists of 10 items, each addressing a specific dimension of functionality or symptoms related to neck disorders.Each item includes five response options ranging from 0 to 5 points, where 0 indicates the absence of problems or limitations and 5 represents the maximum inability or restriction to perform the evaluated activity. The total score is calculated by adding the values of the 10 items, with a maximum of 50 points.

CONTACTS AND LOCATIONS:
Overall Officials: Jasemin Todri, Principal Investigator — UCAM Universidad Catolica San Antonio de Murcia
Locations (1):
- Jasemin Todri, Murcia, Spain